CLINICAL TRIAL: NCT05728216
Title: Histopathological Analysis of Renal Biopsies With Dynamic Full-field Optical Coherence Tomography, a Comparison to Conventional Histopathological Findings for the Diagnosis of Either Acute Kidney Injury or Chronic Kidney Disease in Routine Practices
Brief Title: Histopathological Analysis of Renal Biopsies With Dynamic Full-field Optical Coherence Tomography, a Comparison to Conventional Histopathological Findings for the Diagnosis of Either Acute Kidney Injury or Chronic Kidney Disease in Routine Practices (NEPHROCT)
Acronym: NEPHROCT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier William Morey - Chalon sur Saône (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Thomas Maldiney, Principal Investigator, Centre Hospitalier William Morey - Chalon sur Saône
Other Study IDs: NEPHROCT
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Acute Kidney Injury; Chronic Kidney Diseases; Tomography, Optical Coherence
Keywords: Tomography, Optical Coherence; Chronic Kidney Diseases; Acute Kidney Injury; Kidney Biopsy
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NEPHROCT cohort: Patients > 18 years of age with suspected acute kidney injury or chronic kidney disease requiring biopsy in the nephrology department
  Interventions: Other: Dynamic full-field optical coherence tomography analysis of kidney biopsy

INTERVENTIONS:
Other: Dynamic full-field optical coherence tomography analysis of kidney biopsy — Dynamic full-field optical coherence tomography analysis of kidney biopsy in the nephrology department before conventional histopathological analysis

SUMMARY:
Kidney biopsy play a key role for the investigation of either acute kidney injury or chronic kidney disease. Despite possible complications due to the invasive nature of the biopsy, such procedure is still essential in a number of clinical situations to improve the diagnosis specificity of kidney disease, better inform about its prognosis and guide the management of a future treatment. Pursuing the idea to improve both performance and rapidity associated with the histopathological analysis of kidney biopsy, with a possible recourse to artificial intelligence-based renal pathology, the present study intends to assess the impact of direct histopathological examination of kidney biopsy with dynamic full-field optical coherence tomography in routine practices for the diagnosis of either acute kidney injury or chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years of age with suspected acute kidney injury requiring biopsy in the nephrology department
* patients > 18 years of age with suspected chronic kidney disease requiring biopsy in the nephrology department

Exclusion Criteria:

* inability to perform dynamic full-field optical coherence tomography observation at the moment of kidney biopsy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients > 18 years of age with suspected acute kidney injury or chronic kidney disease requiring biopsy in the nephrology department
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Histopathological analysis of elementary lesions in nephropathology with dynamic full-field optical coherence tomography | Outcome measure is assessed 15 days following kidney biopsy
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify and characterize common glomerular (abnormal / double contour of the glomerular basement membrane, focal segmental glomerulosclerosis, collapse of the glomerular tuft, proliferation of glomerular epithelial cells, endocapillary proliferation, mesangial expansion, necrosis and proliferation with mild increase in extracapillary cells...), vascular (hyaline change, fibrinoid change / necrosis, thrombosis, inflammation or necrosis of vascular walls, arteriosclerosis) and tubulointerstitial (acute tubular necrosis, cytoplasmic vacuolization, lipid inclusions in proximal / distal tubular cells, atrophy of tubules, edema, inflammation or interstitial fibrosis, cortical necrosis) lesions seen in kidney biopsy

SECONDARY OUTCOMES:
Histopathological analysis of healthy kidney biopsy with dynamic full-field optical coherence tomography | Outcome measure is assessed 15 days following kidney biopsy
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify and characterize healthy glomerular (glomerular basement membrane, glomerular tuft, endothelial, epithelial, and mesangial cells, glomerular capsule and capsular space, glomerular capillaries), vascular (afferent and efferent arterioles, interlobular artery) and tubulointerstitial (proximal and distal tubular cells, normal cytoplasmic aspect) structures seen in kidney biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maldiney, Principal Investigator — Centre Hospitalier William Morey - Chalon sur Saône
Locations (1):
- Centre Hospitalier William Morey - Chalon sur Saône, Chalon-sur-Saône, Saône-et-Loire, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hull KL, Adenwalla SF, Topham P, Graham-Brown MP. Indications and considerations for kidney biopsy: an overview of clinical considerations for the non-specialist. Clin Med (Lond). 2022 Jan;22(1):34-40. doi: 10.7861/clinmed.2021-0472. Epub 2021 Dec 17. PMID 34921054
- [Background] Jain M, Robinson BD, Salamoon B, Thouvenin O, Boccara C, Mukherjee S. Rapid evaluation of fresh ex vivo kidney tissue with full-field optical coherence tomography. J Pathol Inform. 2015 Sep 28;6:53. doi: 10.4103/2153-3539.166014. eCollection 2015. PMID 26605118